CLINICAL TRIAL: NCT04053946
Title: Clinical Assessment of the Next Science BlastXTM Antimicrobial Gel and SurgXTM Antimicrobial Gel Healing Efficacy for Below the Knee Amputation Surgical Wound Compared to Standard of Care
Brief Title: Clinical Assessment of Next Science Wound Gels in Healing Below the Knee Amputation Surgical Wound Compared to SOC
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Site backed out
Sponsor: Next Science TM (Industry)
Collaborators: University of Maryland, Baltimore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CSP-012
Record Dates: First submitted 2019-08-09; First posted 2019-08-13 (Actual); Last update posted 2023-04-19 (Actual); Status verified 2023-04

CONDITIONS: Surgical Wound; Surgical Site Infection; Surgical Wound Infection; Amputation Stump; Infection; Surgical Incision
Keywords: BKA; biofilm; Next Science
MeSH Terms: conditions — Surgical Wound; Surgical Wound Infection; Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Next Science (Experimental): Following amputation, SurgX™ will be applied directly to the surgical incision in the operating room under sterile conditions and covered with SOC dressing. The surgical dressing will not be removed until post-operative day 3, except if deemed necessary by the treating surgeon. At that time, direct application of the BlastX™ to the incision will be placed, then covered with a SOC dressing. BlastX™ will be applied every day and covered with SOC dressing.
  Interventions: Device: Next Science Wounds Gels
- Control (No Intervention): Post-op SOC dressing as per treating research doctor to include dressing changes post-op day 3 and daily thereafter.

INTERVENTIONS:
Device: Next Science Wounds Gels — SurgX will be applied once at closure while BlastX will be applied everyday until day 28 with each dressing change.
  Arms: Next Science

SUMMARY:
This is a 64-patient, 90-day, open -label study on adult patients undergoing below knee amputation for various etiologies. The objective of this study is to assess surgical wound healing and wound bioburden using combination treatment of Next Science SurgX™ Antimicrobial Wound Gel and BlastX™ Antimicrobial Wound Gels as compared to standard of care.

DETAILED DESCRIPTION:
This is a prospective, randomized, 90 day, open-label study of patients undergoing below the knee amputation (BKA) with primary closure or completion.

Patients who present for BKA with primary closure or completion will have had a pre-op medical evaluation prior to being screened against the protocol's inclusion/exclusion criteria. If criteria are met, patients will be presented with the option to participate in the study and informed consent procedures will be carried out, in compliance with currently applicable participants' rights and safety regulations.

A minimum of 64 participants, with up to 70 participants, may be enrolled. A participant requiring bilateral BKA will be excluded. Eligible subjects will need to complete the study to meet the primary endpoint.

It is estimated that the study enrollment period will last approximately eighteen months, and the duration of each participants' participation will be three months. Visits in the treatment portion of the study will be carried out at day 0, 3, 14, 21, and 28 days with a scheduling window of 3 days before or after each due date. A phone call follow-up will be conducted at 60 days post-surgery with a window of 7 days before or 14 days after to inquire about the incision (appearance of incision or any noted changes since prior study visit), and overall health of the participant. All participants, regardless of treatment arm, will complete Visit 6 (90 day follow up) with a scheduling window of 7 days before or 21 days after. The key parameters of the study include: percentage of surgical wound area reduction, time patients are deemed ready prosthetic healing, and microorganism type and amounts. Bacterial identification and quantification will occur at days 0, 14, and 28 for all participants.

ELIGIBILITY:
Inclusion Criteria:

1. Male or non-pregnant female 18 years or older
2. Participant must be undergoing below the knee amputation with primary closure or completion below the knee amputation with primary closure.
3. There must be no infection present at the surgical incision site
4. Participant is determined to NOT require endovascular or vascular reconstructive surgery to restore blood flow to the wound within the study period
5. Must have a popliteal pressure on arterial doppler of 40 mm Hg or higher in the surgical leg or angiographic evidence of popliteal artery flow
6. No known allergic reaction or sensitivity to investigational product or components
7. Willing and able to comply with all study procedures including transportation to the study site for all scheduled visits and be available for the duration of the study
8. Provide signed and dated informed consent

Exclusion Criteria:

1. Male or Female less than 18 years old
2. Pregnancy as determined by pre-op urine hCG testing on the day of surgery for women of childbearing potential (women are considered clinically post-menopausal if over 12 consecutive months without a menstrual period)
3. Systemic sepsis at the time of surgery
4. Disseminated Cancer Patients
5. Current long-term (more than 30 consecutive days) use of moderate or high dose oral corticosteroids
6. Current long-term (more than 30 consecutive days) use of immune modulators/suppressors
7. Known sensitivity to investigational product or any components
8. Participants with HIV or acquired immunodeficiency syndrome (AIDS) or any other immunodeficient states
9. Any disease or prior/planned surgery or other situation that in the investigator's opinion may interfere with the participant successfully completing the study.
10. Overlapping participation in another treatment or interventional clinical trial.
11. Family members or students of the Investigator or clinical site.
12. Safety exclusion criterion: At the end of the procedure, the surgeon and PI can discuss to withdraw the patient, if it is felt that continuing in the study will be detrimental to the patient. For example, if the incision cannot be closed, or if it requires a muscle flap, or if the incision site encounters contamination or infection not recognized prior to the start of surgery. The decision to withdraw the patient will be made in the OR, prior to being randomized.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-10-01 (Estimated); Primary Completion 2021-10-01 (Estimated); Study Completion 2021-10-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of Incisional Wound Area Change | 28 Days
  Incisional wounds treated with SurgX™, BlastX™ and SOC Treatment will have higher percentage of area reduction than SOC alone after 28 days of treatment.
Time to when Patient is Ready for Prosthetic Fitting | Day 0 to 90 Days
  Participants treated with SurgX™, BlastX™ and SOC treatment will be deemed ready to be fitted with a prosthetic limb earlier (days) than those in the SOC Control Group.

SECONDARY OUTCOMES:
Bioburden | Day 0, Day 14, Day 28
  The amount of viable microorganisms persisting in wounds (CFU) treated with SurgX™, BlastX™ and SOC treatment will be less than those in the SOC Control Group at one or more of the measured time points.
Bioburden | Day 0, Day 14, Day 28
  The semi-quantitative amount of DNA measured microorganisms persisting in wounds treated with SurgX™, BlastX™ and SOC will be less when compared to the SOC Control Group at one or more of the measured time points.
Bioburden | Day 0, Day 14, Day 28
  The number of DNA measured microorganisms persisting in wounds treated with SurgX™, BlastX™ and SOC treatment will be less when compared to the SOC Control Group at one or more of the measured time points.
Wound Area Reduction | Baseline to 21 days
  Percentage of surgical wound area change after treatment with SurgX™ at the time of the procedure plus 14 and 21 days of treatment with BlastX™ wound gel compared to SOC.

CONTACTS AND LOCATIONS:
Overall Officials: Khanjan H Nagarsheth, MD, MBA, FACS, RPVI, Principal Investigator — University of Maryland

IPD SHARING:
Plan to Share IPD: No